CLINICAL TRIAL: NCT00905619
Title: Functional and Cognitive Impairment in Advanced Kidney Disease
Brief Title: Cognitive Impairment in Kidney Disease
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B5050W-1
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Kidney Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum obtained and kept until end of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control: No kidney disease
- PreHD kidney disease: Kidney disease stage 4 or below
- Hemodialysis: Kidney disease receiving hemodialysis

SUMMARY:
An increasing number of Veterans are anticipated to develop chronic kidney disease (CKD) and require hemodialysis (HD) treatments as the Veteran population ages. In 2003, approximately 290,000 US citizens were receiving HD and an estimated 19 million were affected by CKD. The annual growth rate is predicted to be 7% per year with 500,000 Americans receiving HD treatment by 2010. In 2005, approximately 2500 Veterans were receiving HD with growth expected to parallel that seen in the general population. Whereas Alzheimer's disease is the leading cause of dementia in the general population, growing evidence suggests that patients with advanced CKD experience cognitive deficits related to accelerated cerebrovascular disease. Patients with advanced CKD have been shown to have a high prevalence of sub-clinical cerebrovascular damage on imaging studies and a heavy burden of vascular risk factors such as diabetes, elevated cholesterol, and hypertension. Many of the cognitive deficits related to cerebrovascular disease may go unrecognized by routine measures of cognition. HD patients have increased number of hospitalizations, and several compliance issues ranging from congestive heart failure to dangerous electrolyte imbalances. Impaired cognition in this population is likely to have a significant impact on self-care and compliance with complex medical regimens. Currently, the severity and scope of cognitive impairment related to vascular disease is not well known in patients with advanced kidney disease. Additionally, the relationship between cognitive impairment and measures of self-care independence are not well known. Loss of independence and function secondary to impaired cognitive function is likely to be a significant problem for patients with advanced kidney disease. Early identification of functional impairment, particularly instrumental activities of daily living (IADL), will allow for rehabilitation intervention. Maintaining or improving functional independence through intensive rehabilitation could translate into better compliance and lower hospitalization rate among HD patients. Information obtained from this study is likely to heighten awareness of cognitive impairment and the functional consequences in Veterans with advanced kidney disease. Primary objectives are to determine:

1. The range of cognitive deficits with emphasis on domains affected by vascular disease in patients with advanced CKD and those receiving hemodialysis.
2. The associations between severity of cognitive impairment and severity of kidney disease.
3. The prevalence of impaired IADLs and the level of health-related quality of life (HRQOL) in patients with advanced CKD and those requiring hemodialysis.
4. The relationship or association of cognitive impairment with IADL and HRQOL.

Secondary objective is to determine:

1. The relationships among cerebral and carotid blood flow, carotid artery stiffness, and renal specific metabolic abnormalities with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

PreHD Subjects:

* Male or female with an age of 18 years or older (no upper limit);
* Patients with stage III-IV CKD attending the renal primary care clinic or renal consult clinic;
* Fluent in English;
* Outpatient or stable nursing home patient

HD Subjects:

* Receiving HD for at least two weeks;
* Male or female with an age of 18 years or older (no upper limit);
* Fluent in English;
* Outpatient or stable nursing home patient

Control Subjects:

* Glomerular filtration rate of 60 cc/minute or greater;
* Male or female with an age of 18y or older (no upper limit);
* Fluent in English
* Outpatient

Exclusion Criteria:

PreHD Subjects:

* Acute illness;
* Clinical history of stroke, dementia, or Parkinson's disease;
* Hb <10;
* Liver function tests 2x upper limit of normal;
* Hemodialysis

HD Subjects:

* Acute illness;
* Clinical history of stroke, dementia, or Parkinson's disease;
* Hb <10;
* Liver function tests 2x upper limit of normal;
* URR <65% (measure of dialysis adequacy: will use 3-month average from chart)

Control Subjects:

* Acute illness;
* Clinical history of stroke, dementia, or Parkinson's disease;
* Hb <10;
* Liver function tests 2x upper limit of normal;
* Stage 3-4 CKD;
* Hemodialysis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans at the Bronx VA Renal Clinic, Hemodialysis Unit, and Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2012-09-28 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Assessments | 1 year
  battery of neurocognitive tests

CONTACTS AND LOCATIONS:
Overall Officials: James B Post, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Post JB, Jegede AB, Morin K, Spungen AM, Langhoff E, Sano M. Cognitive profile of chronic kidney disease and hemodialysis patients without dementia. Nephron Clin Pract. 2010;116(3):c247-55. doi: 10.1159/000317206. Epub 2010 Jul 2. PMID 20606486
- [Result] Post JB, Morin KG, Handrakis JP, Rivera DR, Yen C, Sano M, Spungen AM. Cognition may be related to arterial pulsatility index in HD patients. Clin Nephrol. 2014 May;81(5):313-9. doi: 10.5414/cn107998. PMID 24780553